CLINICAL TRIAL: NCT03842631
Title: Optimizing Timolol Maleate Treatment of Infantile Hemangioma by Doppler Ultrasound Examination: a Single Center, Open Cohort Study.
Brief Title: Optimizing Timolol Maleate Treatment of Infantile Hemangioma by Doppler Ultrasound Examination
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: XiaoXi Lin (Other)
Responsible Party: Sponsor-Investigator, XiaoXi Lin, Professor, Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University
Organization: Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University (Other)
Other Study IDs: SH9H-2018-T48-2
Record Dates: First submitted 2019-02-02; First posted 2019-02-15 (Actual); Last update posted 2019-02-19 (Actual); Status verified 2019-02

CONDITIONS: Infantile Hemangioma
Keywords: Timolol Maleate; Doppler Ultrasound Examination
MeSH Terms: conditions — Hemangioma, Capillary | interventions — Timolol

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Superficial Group: Hemangioma depth evaluated by B-ultrasonoscope is lower than or equal to 6mm. After enrollment, patients would be subject to external use of Timolol Maleate 0.5% Oph Soln for the treatment of hemangioma.
  Interventions: Drug: Timolol Maleate 0.5% Oph Soln
- Deep Group: Hemangioma depth evaluated by B-ultrasonoscope is more than 6mm. After enrollment, patients would be subject to external use of Timolol Maleate 0.5% Oph Soln for the treatment of hemangioma.
  Interventions: Drug: Timolol Maleate 0.5% Oph Soln

INTERVENTIONS:
Drug: Timolol Maleate 0.5% Oph Soln — External use of 0.5% Timolol Maleate Drops for all patients in different depths of IH lesion.
  Other Names: 0.5% Timolol Maleate Drops

SUMMARY:
The purpose of this study is to assess the safety and efficacy of Timolol Maleate treatment for different depth of infantile hemangioma based on B-ultrasonography. Based on the depth of hemangioma, patients will be proactively allocated to two groups. And then, all patients in both groups will receive topical timolol treatment in the same protocol and dosage.

DETAILED DESCRIPTION:
Primary: Describe the efficacy of 0.5% topical timolol maleate drops in different depth of infantile hemangioma as assessed through IB-ultrasound.

ELIGIBILITY:
Inclusion Criteria:

* Infants of 0 to 6 months of age
* Skin Infantile hemangiomas (IHs) in the proliferation stage without prior treatment
* IHs with a surface area of less than 1% of body surface area
* Skin type III/IV

Exclusion Criteria:

* Ulcerated IHs.
* Unsuitable for topical Timolol treatment due to anatomical location of lesion, eg.

periorbital and lip IHs.

* Patients with severe systemic or congenital disease which may affect the patient's safety in this study

Max Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Patients with infantile hemangiomas presented to the outpatient clinic of Shanghai Ninth People's Hospital would be considered for enrolment in the study. The diagnosis of proliferating infantile hemangioma is based on medical history and B-ultrasonography.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2019-02-16 (Actual); Primary Completion 2020-06-01 (Estimated); Study Completion 2020-12-01 (Estimated)

PRIMARY OUTCOMES:
Depth of infantile hemangioma | through study completion, an average of 1 year
  At the beginning of treatment, the thickness of hemangioma was measured by b-mode ultrasound at each follow-up.

SECONDARY OUTCOMES:
Color | through study completion, an average of 1 year
  The redness of lesion is measured by standard photography.
Dimensions | through study completion, an average of 1 year
  The dimension of lesion is measured by standard photography.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoxi Lin, PhD, Principal Investigator — Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University
Locations (1):
- Shanghai Ninth People's hospital, Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided